CLINICAL TRIAL: NCT04456777
Title: Effect of Vortioxetine on Cognitive Symptoms in Patients With
Brief Title: Effect of Vortioxetine on Cognitive Symptoms in Patients With Schizophrenia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alen Greš (Other)
Responsible Party: Sponsor-Investigator, Alen Greš, Alen Greš,MD, Clinical Hospital Centre Zagreb
Organization: Clinical Hospital Centre Zagreb (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: evcps
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Cognitive Deficit
MeSH Terms: conditions — Cognition Disorders | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1group (Experimental): patients with vortioxetine
  Interventions: Drug: Vortioxetine
- 2 group (Placebo Comparator): patients without vortioxetine
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — vortioxetine will be administreted for 3 months

SUMMARY:
Research goals:

1. Examination of the relationship between the use of vortioxetine and cognitive efficacy in patients with schizophrenia.
2. Examination of the association between the use of vortioxetine and the presence depressive symptoms, physical and social anhedonia in patients with the disease from schizophrenia.
3. Examining the association between vortioxetine use and quality of life

(functional recovery) in patients with schizophrenia

Expected results (hypotheses)

1. Patients with schizophrenia treated with additional therapy vortioxetine will show better cognitive achievement in memory (short-term and long-term), attention, logical reasoning and reasoning, speed of information processing, processing of visual and sound information, language and speech in relation to patients without additional intervention.
2. Patients with schizophrenia treated with additional therapy vortioxetine will have a less pronounced presence of depressive symptoms, physical and social anhedonia in relation to untreated patients with additional vortioxetine therapy.
3. Patients with schizophrenia who were treated with additional therapy vortioxetine will have a better quality of life, ie. better functional recovery

DETAILED DESCRIPTION:
In the first phase of the research, the development of the research protocol and obtaining it will be done of his approval.

The second phase of the research will include patients with schizophrenia disorders based on inclusive and exclusive criteria and a study will be conducted procedure. In the third phase of the research, the obtained results are processed and analyzed.

The content of the dissertation will include an introduction, a goal with hypotheses, methods, results, discussion, conclusions and literature. In the introduction, in addition to current knowledge about schizophrenia and vortioxetine, it will be pointed out cognition problem in patients with schizophrenia.

It will be defined and explained hypotheses and research objectives. In the chapter dedicated to methodology, the number of respondents and a description will be presented study concepts, presentation of statistical methods used for data processing The presentation of the results obtained by this study will be presented textually, tabularly and using charts. The obtained results will be commented and evaluated in the Discussion. Recent literature will be used

Randomization 1:1 will divide 120 patients with schizophrenia into two groups, each group into 3 subgroups. One group of 60 patients (who are on monotherapy antipsychotics: new generations: 20 patients will be on olanzapine, 20 patients on risperidone and 20 patients on aripiprazole) will receive vortioxetine and the other control group of 60 patients (who is also on monotherapy with new antipsychotics generations: 20 patients will be on olanzapine, 20 patients on risperidone and 20 patients on aripiprazole) will not receive vortioxetine. Vortioxetine will be given in 10 mg dose (which can be reduced by 5 mg if needed in case of poor tolerability)

1. Initial examination:

   International mini neuropsychiatric interview (M.I.N.I.) publicly available, works doctor General questionnaire - designed by a doctor Positive and negative syndrome scales (PANSS) are publicly available, by a doctor The Calgary Depression Scale for Schizophrenia (CDSS) is publicly available, it works doctor World Health Organization for Quality of Life (WHOQOL-BREF) publicly available, works doctor Chapman (social anhedonia and physical anhedonia) - publicly available, works doctor Wechsler WAIS IV (subtests: numerical memory test; encryption test symbols) - available at Naklada Slap, Zagreb, HR, by a clinical psychologist

   Screening tests:
   1. Mini-mental state (MMSE) or Folstein test - publicly available, by a doctor
   2. Montreal Cognitive Assessment (MoCA) - publicly available, by a physician
2. At the end of the second month:

   International mini neuropsychiatric interview (M.I.N.I.) publicly available, works doctor Mini-mental state (MMSE) or Folstein test - publicly available, by a doctor Montreal Cognitive Assessment (MoCA) - publicly available, by a doctor
3. At the end of the third month:

International mini neuropsychiatric interview (M.I.N.I.) publicly available, works doctor Positive and negative syndrome scales (PANSS) are publicly available, by a doctor The Calgary Depression Scale for Schizophrenia (CDSS) is publicly available, it works doctor World Health Organization for Quality of Life (WHOQOL-BREF) publicly available, works doctor Chapman (social anhedonia and physical anhedonia) - publicly available, works doctor Wechsler WAIS IV (subtests: numerical memory test; encryption test)

- Available at Naklada Slap, Zagreb, HR, by a clinical psychologist Screening tests: a) Mini-mental state (MMSE) or Folstein test - public

available, works doctor b) Montreal Cognitive Assessment (MoCA) - publicly available, by a doctor It is expected: improvement of cognitive functions in relation to the initial examination

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50, informed consent signed, confirmed diagnosis of schizophrenia, taking monotherapy with antipsychotics: aripiprazole, risperidone, paliperidone or olanzapine, unchanged dose maintenance back at least 6 months, remission of psychotic symptoms (PANSS ≤ 70), and that they do not have any of the exclusive criteria:

Exclusion Criteria:

* taking benzodiazepines at doses equivalent to ≥ 10 mg diazepam, taking mood stabilizers, antidepressants three months ago, abuse of addictions back three months, suicide attempt back 6 months, suicidal, heteroaggressive, or other similar behavior back 6 months, somatic comorbidities affecting cognitive functions (intellectual disabilities, significant neurological disease or head trauma), pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
better cognitive functions | 2 years
  improvement of cognitive functions compared to initial examination

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Centre Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No